CLINICAL TRIAL: NCT01426386
Title: A Randomised, Controlled, Assessor-blind, Parallel Groups, Multi-national, Multi-centre Trial Assessing the Dose-response Relationship of FE 999049 in Controlled Ovarian Stimulation in Women Undergoing an ART Programme
Brief Title: A Dose-response Trial Using rFSH FE 999049 in Women Undergoing IVF/ICSI Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 000009; 2011-000633-36 (EudraCT Number)
Record Dates: First submitted 2011-08-30; First posted 2011-08-31 (Estimated); Results first posted 2018-08-03 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2018-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — FE 999049; Glycoprotein Hormones, alpha Subunit

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 5.2 µg (Experimental)
  Interventions: Drug: FE 999049
- 6.9 µg (Experimental)
  Interventions: Drug: FE 999049
- 8.6 µg (Experimental)
  Interventions: Drug: FE 999049
- 10.3 µg (Experimental)
  Interventions: Drug: FE 999049
- 12.1 µg (Experimental)
  Interventions: Drug: FE 999049
- 11 µg FbM (150 IU) (Active Comparator)
  Interventions: Drug: Gonal - F

INTERVENTIONS:
Drug: FE 999049
  Arms: 10.3 µg; 12.1 µg; 5.2 µg; 6.9 µg; 8.6 µg
Drug: Gonal - F
  Arms: 11 µg FbM (150 IU)

SUMMARY:
This trial investigates the effects of several doses of FE 999049 in women undergoing IVF/ICSI (in-vitro fertilisation/intracytoplasmic sperm injection) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with tubal infertility, unexplained infertility, infertility related to endometriosis stage I/II or with partners diagnosed with male factor infertility
* Women eligible for IVF (in-vitro fertilisation) and/or ICSI (intracytoplasmic sperm injection) treatment
* Women aged 18-37 years
* Women with body mass index (BMI) of 18.5-32.0 kg/m2

Exclusion Criteria:

* Women with polycystic ovary syndrome (PCOS) associated with anovulation, endometriosis stage III/IV
* Women with history of recurrent miscarriage
* Women with contraindications to controlled ovarian stimulation with gonadotropins
* Women with three or more controlled ovarian stimulation cycles

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 265 (Actual)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (8):
- Belgium (2):
  - UZ Brussel, Brussels
  - UZ Gent, Ghent
- ICF CUBE, Prague, Czechia
- Rigshospitalet, Copenhagen, Denmark
- Spain (4):
  - IU Dexeus, Barcelona
  - IVI Madrid, Madrid
  - IVI Sevilla, Seville
  - IVI Valencia, Valencia

REFERENCES:
- [Result] Arce JC, Larsson P, Garcia-Velasco JA. Establishing the follitropin delta dose that provides a comparable ovarian response to 150 IU/day follitropin alfa. Reprod Biomed Online. 2020 Oct;41(4):616-622. doi: 10.1016/j.rbmo.2020.07.006. Epub 2020 Jul 15. PMID 32819842
- [Derived] Arce JC, Andersen AN, Fernandez-Sanchez M, Visnova H, Bosch E, Garcia-Velasco JA, Barri P, de Sutter P, Klein BM, Fauser BC. Ovarian response to recombinant human follicle-stimulating hormone: a randomized, antimullerian hormone-stratified, dose-response trial in women undergoing in vitro fertilization/intracytoplasmic sperm injection. Fertil Steril. 2014 Dec;102(6):1633-40.e5. doi: 10.1016/j.fertnstert.2014.08.013. Epub 2014 Sep 23. PMID 25256937

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 7 sites randomised subjects to the trial: 1 in Belgium, 1 in Czech Republic, 1 in Denmark and 4 in Spain.
Pre-assignment Details: In total 334 subjects were screened. Of these, 69 were screening failures and 265 were randomised. All randomised subjects were exposed to investigational medicinal product (IMP).
Groups:
- FE 999049 5.2 µg: Subjects received single daily subcutaneous injections of 5.2 µg FE 999049, for a maximum of 16 days
- FE 999049 6.9 µg: Subjects received single daily subcutaneous injections of 6.9 µg FE 999049, for a maximum of 16 days
- FE 999049 8.6 µg: Subjects received single daily subcutaneous injections of 8.6 µg FE 999049, for a maximum of 16 days
- FE 999049 10.3 µg: Subjects received single daily subcutaneous injections of 10.3 µg FE 999049, for a maximum of 16 days
- FE 999049 12.1 µg: Subjects received single daily subcutaneous injections of 12.1 µg FE 999049, for a maximum of 16 days
- GONAL-F 11 µg: Subjects received single daily subcutaneous injections of 11 µg GONAL-F, for a maximum of 16 days
Period: Overall Study
Arm/Group | FE 999049 5.2 µg | FE 999049 6.9 µg | FE 999049 8.6 µg | FE 999049 10.3 µg | FE 999049 12.1 µg | GONAL-F 11 µg
Started | 42 | 45 | 44 | 44 | 47 | 43
Completed | 39 | 39 | 42 | 44 | 43 | 42
Not Completed | 3 | 6 | 2 | 0 | 4 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Did not attend scheduled visit | 1 | 4 | 0 | 0 | 2 | 1
Not completed — Poor response | 2 | 1 | 2 | 0 | 1 | 0
Not completed — Personal reasons | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FE 999049 5.2 µg | FE 999049 6.9 µg | FE 999049 8.6 µg | FE 999049 10.3 µg | FE 999049 12.1 µg | GONAL-F 11 µg | Total
Number analyzed (Participants) | 42 | 45 | 44 | 44 | 47 | 43 | 265
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (2.24) | 32.3 (3.51) | 32.8 (2.44) | 32.3 (3.21) | 32.6 (2.97) | 32.4 (3.04) | 32.7 (2.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 45 | 44 | 44 | 47 | 43 | 265
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Oocytes Retrieved
Time Frame: Day of oocyte retrieval (up to Day 18 after start of stimulation)
Population: Modified Intention-to-treat (mITT) population (all randomised and exposed subjects). This is equivalent to the Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Oocytes
Arm/Group | FE 999049 5.2 µg | FE 999049 6.9 µg | FE 999049 8.6 µg | FE 999049 10.3 µg | FE 999049 12.1 µg | GONAL-F 11 µg
Number analyzed (Participants) | 42 | 45 | 44 | 44 | 47 | 43
Oocytes | 5.2 (3.3) | 7.9 (5.9) | 9.2 (4.6) | 10.5 (7.0) | 12.2 (5.9) | 10.4 (5.2)
Statistical Analysis 1: Comparison: FE 999049 5.2 µg vs FE 999049 6.9 µg vs FE 999049 8.6 µg vs FE 999049 10.3 µg vs FE 999049 12.1 µg; The dose-response relationship was analysed using an analysis of covariance (ANCOVA) model; Test type: Other — Based on the ANCOVA model the slope of the dose-response curve was estimated. Null hypothesis: Slope of dose-response curve equal to 0 (zero); p < 0.001, ANCOVA — The a priori threshold for statistical significance was 5% (two-sided); Number of oocytes retrieved as dependent variable, centre and AMH strata (5.0-14.9 pmol/L and 15.0-44.9 pmol/L) as factors and log(dose) as covariate; Slope of the dose-response curve = 7.9, 95% CI 2-sided [5.69 to 10.18]

2. Secondary Outcome: Number and Size of Follicles During Stimulation
Description: Follicular volume at end of stimulation
Time Frame: End of stimulation (up to 16 stimulation days)
Population: mITT population (all randomised and exposed subjects). This is equivalent to the FAS
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | FE 999049 5.2 µg | FE 999049 6.9 µg | FE 999049 8.6 µg | FE 999049 10.3 µg | FE 999049 12.1 µg | GONAL-F 11 µg
Number analyzed (Participants) | 42 | 45 | 44 | 44 | 47 | 43
cm^3 | 19.2 (7.0) | 23.0 (10.5) | 25.0 (9.2) | 27.9 (15.6) | 28.2 (9.5) | 26.7 (9.2)
Statistical Analysis 1: Comparison: FE 999049 5.2 µg vs FE 999049 6.9 µg vs FE 999049 8.6 µg vs FE 999049 10.3 µg vs FE 999049 12.1 µg; The dose-response relationship was analysed using an analysis of covariance (ANCOVA) model; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA — No adjustment for multiplicity was applied for the secondary endpoints; Follicular volume as dependent variable, centre and AMH strata (5.0-14.9 pmol/L and 15.0-44.9 pmol/L) as factors and log(dose) as covariate; Slope of the dose-response curve = 11.1, 95% CI 2-sided [6.78 to 15.48]

3. Secondary Outcome: Endocrine Profile
Description: Estradiol at end of stimulation
Time Frame: End of stimulation (up to 16 stimulation days)
Population: mITT population (all randomised and exposed subjects). This is equivalent to the FAS
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | FE 999049 5.2 µg | FE 999049 6.9 µg | FE 999049 8.6 µg | FE 999049 10.3 µg | FE 999049 12.1 µg | GONAL-F 11 µg
Number analyzed (Participants) | 42 | 45 | 44 | 44 | 47 | 43
pmol/L | 3641.9 (2954.6) | 5221.1 (3378.8) | 5689.5 (3995.7) | 6171.8 (3855.9) | 6442.0 (3195.2) | 5750.7 (3709.7)
Statistical Analysis 1: Comparison: FE 999049 5.2 µg vs FE 999049 6.9 µg vs FE 999049 8.6 µg vs FE 999049 10.3 µg vs FE 999049 12.1 µg; The dose-response relationship was analysed using an analysis of covariance (ANCOVA) model; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA — No adjustment for multiplicity was applied for the secondary endpoints; Log(estradiol) as dependent variable, AMH strata (5.0-14.9 pmol/L and 15.0-44.9 pmol/L) as factor, log(dose) and log(baseline estradiol) as covariates; Slope of the dose-response curve = 0.8, 95% CI 2-sided [0.56 to 1.11]

4. Secondary Outcome: Total IMP Dose
Time Frame: End of stimulation (up to 16 stimulation days)
Population: mITT population (all randomised and exposed subjects). This is equivalent to the FAS
Measure: Mean (Standard Deviation); unit: µg
Arm/Group | FE 999049 5.2 µg | FE 999049 6.9 µg | FE 999049 8.6 µg | FE 999049 10.3 µg | FE 999049 12.1 µg | GONAL-F 11 µg
Number analyzed (Participants) | 42 | 45 | 44 | 44 | 47 | 43
µg | 50.0 (11.6) | 61.9 (13.7) | 71.9 (14.1) | 81.0 (14.2) | 97.8 (22.0) | 94.7 (18.1)

5. Secondary Outcome: Number of Fertilised Oocytes
Description: An oocyte with 2 pronuclei was regarded as correctly fertilised
Time Frame: Day 1 after insemination
Population: Subjects with oocytes retrieved
Measure: Mean (Standard Deviation); unit: Fertilised oocytes
Arm/Group | FE 999049 5.2 µg | FE 999049 6.9 µg | FE 999049 8.6 µg | FE 999049 10.3 µg | FE 999049 12.1 µg | GONAL-F 11 µg
Number analyzed (Participants) | 42 | 45 | 44 | 44 | 47 | 43
Fertilised oocytes | 3.7 (2.5) | 5.4 (3.8) | 4.9 (2.7) | 6.1 (5.1) | 6.7 (3.5) | 6.4 (3.5)
Statistical Analysis 1: Comparison: FE 999049 5.2 µg vs FE 999049 6.9 µg vs FE 999049 8.6 µg vs FE 999049 10.3 µg vs FE 999049 12.1 µg; The dose-response relationship was analysed using an analysis of covariance (ANCOVA) model; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA — No adjustment for multiplicity was applied for the secondary endpoints; Fertilised oocytes as dependent variable, AMH strata (5.0-14.9 pmol/L and 15.0-44.9 pmol/L) as factor and log(dose) as covariate; Slope of the dose-response curve = 3.2, 95% CI 2-sided [1.71 to 4.78]

6. Secondary Outcome: Number and Quality of Blastocysts on Day 5
Description: Number of blastocysts (total and good-quality) on Day 5 are presented. A good-quality blastocyst was defined as a blastocyst of grade 3BB or higher
Time Frame: Day 5 after oocyte retrieval
Population: Subjects with oocytes retrieved
Measure: Mean (Standard Deviation); unit: Blastocysts
Arm/Group | FE 999049 5.2 µg | FE 999049 6.9 µg | FE 999049 8.6 µg | FE 999049 10.3 µg | FE 999049 12.1 µg | GONAL-F 11 µg
Number analyzed (Participants) | 42 | 45 | 44 | 44 | 47 | 43
Blastocysts
  Total blastocysts | 2.3 (1.7) | 3.1 (2.7) | 2.7 (2.0) | 2.8 (2.8) | 3.2 (2.2) | 3.5 (2.5)
  Good quality blastocysts | 0.9 (1.2) | 1.4 (1.7) | 1.2 (1.2) | 1.4 (1.5) | 1.3 (1.3) | 1.6 (1.6)

7. Secondary Outcome: Clinical Pregnancy With Fetal Heart Beat Rate
Description: Clinical pregnancy with fetal heart beat was defined as at least one intrauterine gestational sac with fetal heart beat
Time Frame: 5-6 weeks after transfer
Population: mITT population (all randomised and exposed subjects). This is equivalent to the FAS
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | FE 999049 5.2 µg | FE 999049 6.9 µg | FE 999049 8.6 µg | FE 999049 10.3 µg | FE 999049 12.1 µg | GONAL-F 11 µg
Number analyzed (Participants) | 42 | 45 | 44 | 44 | 47 | 43
percentage | 36 [21.6 to 52.0] | 40 [25.7 to 55.7] | 36 [22.4 to 52.2] | 25 [13.2 to 40.3] | 40 [26.4 to 55.7] | 51 [35.5 to 66.7]
Statistical Analysis 1: Comparison: FE 999049 5.2 µg vs FE 999049 6.9 µg vs FE 999049 8.6 µg vs FE 999049 10.3 µg vs FE 999049 12.1 µg vs GONAL-F 11 µg; Test type: Other — Treatment groups were compared using the chi-squared test; p = 0.248, Chi-squared — No adjustment for multiplicity was applied for the secondary endpoints

8. Secondary Outcome: Frequency and Intensity of Adverse Events
Time Frame: From signing informed consent form until end of trial visit (up to 5 months)
Population: Safety population (all randomised and exposed subjects). This is equivalent to the mITT
Measure: Number; unit: participants
Arm/Group | FE 999049 5.2 µg | FE 999049 6.9 µg | FE 999049 8.6 µg | FE 999049 10.3 µg | FE 999049 12.1 µg | GONAL-F 11 µg
Number analyzed (Participants) | 42 | 45 | 44 | 44 | 47 | 43
participants
  Any mild adverse events | 15 | 17 | 17 | 18 | 15 | 11
  Any moderate adverse events | 2 | 6 | 5 | 9 | 8 | 2
  Any severe adverse events | 0 | 0 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: From signing informed consent form until the end of trial visit (up to 5 months)
Arm/Group | FE 999049 5.2 µg | FE 999049 6.9 µg | FE 999049 8.6 µg | FE 999049 10.3 µg | FE 999049 12.1 µg | GONAL-F 11 µg
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/45 | 0/44 | 0/44 | 0/47 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/45 | 0/44 | 1/44 | 0/47 | 0/43
Other Adverse Events (participants affected / at risk) | 11/42 | 9/45 | 11/44 | 12/44 | 11/47 | 4/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FE 999049 5.2 µg (N=42) | FE 999049 6.9 µg (N=45) | FE 999049 8.6 µg (N=44) | FE 999049 10.3 µg (N=44) | FE 999049 12.1 µg (N=47) | GONAL-F 11 µg (N=43)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FE 999049 5.2 µg (N=42) | FE 999049 6.9 µg (N=45) | FE 999049 8.6 µg (N=44) | FE 999049 10.3 µg (N=44) | FE 999049 12.1 µg (N=47) | GONAL-F 11 µg (N=43)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 4 (4) | 5 (5) | 3 (4) | 1 (1) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 5 (5) | 2 (2) | 5 (5) | 5 (5) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 4 (4) | 3 (4) | 2 (2) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.